CLINICAL TRIAL: NCT03259269
Title: endTB (Expand New Drugs for TB) Observational Study: Treatment of MDR-TB With Regimens Containing Bedaquiline or Delamanid
Brief Title: Expand New Drugs for TB [endTB]
Status: Completed | Type: Observational
Sponsor: Partners in Health (Other)
Collaborators: Médecins Sans Frontières, France (Other); Interactive Research and Development (Other); Harvard Medical School (HMS and HSDM) (Other); Epicentre (Other)
Responsible Party: Sponsor
Other Study IDs: Partners IRB 2015P001669
Record Dates: First submitted 2017-08-21; First posted 2017-08-23 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2022-06

CONDITIONS: Tuberculosis, Multidrug-Resistant
MeSH Terms: conditions — Tuberculosis, Multidrug-Resistant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Bedaquiline and companion WHO Group 5 drugs
  Interventions: Other: This is a non-intervention observational study
- Delamanid and companion WHO Group 5 drugs
  Interventions: Other: This is a non-intervention observational study

INTERVENTIONS:
Other: This is a non-intervention observational study — No applicable intervention; this is a secondary data analysis observational study.

SUMMARY:
This observational study will examine the safety and efficacy of bedaquiline and delamanid used (individually, not together) in routine, multidrug regimens for treatment of MDR-TB. The information gathered in this study will inform doctors how best to use these TB drugs in the future.

ELIGIBILITY:
Inclusion Criteria:

* Any patient who receives a treatment regimen containing bedaquiline or delamanid at an endTB site will be invited to participate in this observational study, regardless of age or gender.
* Any patient who signs the study informed consent form will be included in the study.

Exclusion Criteria:

* Refusal to participate in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All MDR-TB patients started on treatment containing a new TB drug (bedaquiline or delamanid) and enrolled in clinical care within the endTB Project.
Sampling Method: Non-Probability Sample
Enrollment: 2804 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
End of treatment outcome | 20 - 24 months of treatment
  Final outcomes: cured, treatment completed, treatment failed, lost to follow-up, died, not evaluated

CONTACTS AND LOCATIONS:
Locations (16):
- National Treatment Centre for Tuberculosis, Abovian, Armenia, Abovyan, Armenia
- National Institute of Diseases of the Chest and Hospital (NIDCH), Dhaka, Dhaka, Bangladesh
- Republican Research and Practical Centre for Pulmonology and Tuberculosis, Minsk, Belarus
- Aung San Tuberculosis Hospital, Yangon, Burma
- Bishoftu Hospital, Bishoftu, Ethiopia
- National Center for Tuberculosis and Lung Diseases, Tbilisi, Georgia
- RS Islam Jakarta Cempaka Putih, Jakarta, Indonesia
- National Research Center for Phthisionpulmonology, Almaty, Kazakhstan
- MSF Tuberculosis clinic, Mathare, Nairobi, Kenya, Nairobi, Kenya
- Kara-Suu District TB hospital, Kara Suu, Kyrgyzstan
- Botshabelo Hospital, Maseru, Lesotho
- Pakistan (3):
  - The Indus Hospital, Karachi, Karachi
  - Institute of Chest Diseases, Kotri, Kotri
  - Gulab Devi Chest Hospital, Lahore, Lahore
- Socios en Salud, Carabayllo, Peru
- King Dinuzulu Hospital, Durban, South Africa

REFERENCES:
- [Background] Huerga H, Khan U, Bastard M, Mitnick CD, Lachenal N, Khan PY, Seung KJ, Melikyan N, Ahmed S, Rich ML, Varaine F, Osso E, Rashitov M, Salahuddin N, Salia G, Sanchez E, Serobyan A, Rafi Siddiqui M, Grium Tefera D, Vetushko D, Yeghiazaryan L, Holtzman D, Islam S, Kumsa A, Jacques Leblanc G, Leonovich O, Mamsa S, Manzur-Ul-Alam M, Myint Z, Padayachee S, Franke MF, Hewison C. Safety and Effectiveness Outcomes From a 14-Country Cohort of Patients With Multi-Drug Resistant Tuberculosis Treated Concomitantly With Bedaquiline, Delamanid, and Other Second-Line Drugs. Clin Infect Dis. 2022 Oct 12;75(8):1307-1314. doi: 10.1093/cid/ciac176. PMID 35243494
- [Background] Hewison C, Khan U, Bastard M, Lachenal N, Coutisson S, Osso E, Ahmed S, Khan P, Franke MF, Rich ML, Varaine F, Melikyan N, Seung KJ, Adenov M, Adnan S, Danielyan N, Islam S, Janmohamed A, Karakozian H, Kamene Kimenye M, Kirakosyan O, Kholikulov B, Krisnanda A, Kumsa A, Leblanc G, Lecca L, Nkuebe M, Mamsa S, Padayachee S, Thit P, Mitnick CD, Huerga H. Safety of Treatment Regimens Containing Bedaquiline and Delamanid in the endTB Cohort. Clin Infect Dis. 2022 Sep 29;75(6):1006-1013. doi: 10.1093/cid/ciac019. PMID 35028659
- [Background] Khan PY, Franke MF, Hewison C, Seung KJ, Huerga H, Atwood S, Ahmed S, Khan M, Sultana T, Manzur-Ul-Alam M, Vo LNQ, Lecca L, Yae K, Kozhabekov S, Tamirat M, Gelin A, Vilbrun SC, Kikvidze M, Faqirzai J, Kadyrov A, Skrahina A, Mesic A, Avagyan N, Bastard M, Rich ML, Khan U, Mitnick CD. All-oral longer regimens are effective for the management of multidrug-resistant tuberculosis in high-burden settings. Eur Respir J. 2022 Jan 20;59(1):2004345. doi: 10.1183/13993003.04345-2020. Print 2022 Jan. PMID 34140298
- [Background] Maretbayeva SM, Rakisheva AS, Adenov MM, Yeraliyeva LT, Algozhin YZ, Stambekova AT, Berikova EA, Yedilbayev A, Rich ML, Seung KJ, Issayeva AM. Culture conversion at six months in patients receiving bedaquiline- and delamanid-containing regimens for the treatment of multidrug-resistant tuberculosis. Int J Infect Dis. 2021 Dec;113 Suppl 1:S91-S95. doi: 10.1016/j.ijid.2021.03.075. Epub 2021 Apr 3. PMID 33823277
- [Background] Franke MF, Khan P, Hewison C, Khan U, Huerga H, Seung KJ, Rich ML, Zarli K, Samieva N, Oyewusi L, Nair P, Mudassar M, Melikyan N, Lenggogeni P, Lecca L, Kumsa A, Khan M, Islam S, Hussein K, Docteur W, Chumburidze N, Berikova E, Atshemyan H, Atwood S, Alam M, Ahmed S, Bastard M, Mitnick CD. Culture Conversion in Patients Treated with Bedaquiline and/or Delamanid. A Prospective Multicountry Study. Am J Respir Crit Care Med. 2021 Jan 1;203(1):111-119. doi: 10.1164/rccm.202001-0135OC. PMID 32706644
- [Background] Seung KJ, Franke MF, Hewison C, Huerga H, Khan U, Mitnick CD; end TB Study Group. High prevalence of hepatitis C infection among multidrug-resistant tuberculosis patients. J Hepatol. 2020 May;72(5):1028-1029. doi: 10.1016/j.jhep.2019.10.018. Epub 2020 Mar 6. No abstract available. PMID 32147086
- [Background] Seung KJ, Khan P, Franke MF, Ahmed S, Aiylchiev S, Alam M, Putri FA, Bastard M, Docteur W, Gottlieb G, Hewison C, Islam S, Khachatryan N, Kotrikadze T, Khan U, Kumsa A, Lecca L, Tassew YM, Melikyan N, Naing YY, Oyewusi L, Rich M, Wanjala S, Yedilbayev A, Huerga H, Mitnick CD. Culture Conversion at 6 Months in Patients Receiving Delamanid-containing Regimens for the Treatment of Multidrug-resistant Tuberculosis. Clin Infect Dis. 2020 Jul 11;71(2):415-418. doi: 10.1093/cid/ciz1084. PMID 31676905
- [Background] Khan U, Huerga H, Khan AJ, Mitnick CD, Hewison C, Varaine F, Bastard M, Rich M, Franke MF, Atwood S, Khan PY, Seung KJ. The endTB observational study protocol: treatment of MDR-TB with bedaquiline or delamanid containing regimens. BMC Infect Dis. 2019 Aug 20;19(1):733. doi: 10.1186/s12879-019-4378-4. PMID 31429722
- [Background] Lachenal N, Hewison C, Mitnick C, Lomtadze N, Coutisson S, Osso E, Ahmed S, Leblanc G, Islam S, Atshemyan H, Nair P, Kholikulov B, Aiylchiev S, Zarli K, Adnan S, Krisnanda A, Padayachee S, Stambekova A, Sahabutdinova Y, de Guadalupe S, Moreno P, Kumsa A, Reshid A, Makaka J, Abebe S, Melikyan N, Seung KJ, Khan U, Khan P, Huerga H, Rich M, Varaine F. Setting up pharmacovigilance based on available endTB Project data for bedaquiline. Int J Tuberc Lung Dis. 2020 Oct 1;24(10):1087-1094. doi: 10.5588/ijtld.20.0115. PMID 33126944
- [Background] Seung KJ, Khan U, Varaine F, Ahmed S, Bastard M, Cloez S, Damtew D, Franke MF, Herboczek K, Huerga H, Islam S, Karakozian H, Khachatryan N, Kliesckova J, Khan AJ, Khan M, Khan P, Kotrikadze T, Lachenal N, Lecca L, Lenggogeni P, Maretbayeva S, Melikyan N, Mesic A, Mitnick CD, Mofolo M, Perrin C, Richard M, Tassew YM, Telnov A, Vilbrun SC, Wanjala S, Rich ML, Hewison C. Introducing new and repurposed TB drugs: the endTB experience. Int J Tuberc Lung Dis. 2020 Oct 1;24(10):1081-1086. doi: 10.5588/ijtld.20.0141. PMID 33126943
- See also: endTB Project website — http://endtb.org/